CLINICAL TRIAL: NCT04495504
Title: The Effect of Continuous Administration of Ropivacaine by Bi-laterosternal Multiperforated Catheters Placed Before a Sternotomy for Cardiac Surgery
Brief Title: Administration of Ropivacaine by Bi-laterosternal Multiperforated Catheters Placed Before a Sternotomy for Cardiac Surgery
Acronym: Pre-BLS-Sterno
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pré-BLS-Sterno-RBHP 2018 ELJEZ
Record Dates: First submitted 2020-07-23; First posted 2020-08-03 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Scheduled Cardiac Surgery; Age Under 85 Years
Keywords: Postoperative analgesia; Sternotomy; Local anesthetics
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: Placement by the surgeon of two catheters in BLS position before the surgical incision. Administration of a bolus dose of 10 ml of ropivacaine 7, 5 mg/mL in each catheter followed by a continuous infusion of ropivacaine 2 mg/ml in a rate of 3 mL/h during the first 48 hours postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ropivacaine group (Experimental): Administration of a bolus dose of ropivacaine, followed by a continuous infusion of ropivacaine during the first 48 hours postoperatively.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — Administration of a bolus dose of 10 ml of ropivacaine 7, 5 mg/mL in each catheter Continuous infusion of ropivacaine 2 mg/ml in a rate of 3 mL/h during the first 48 hours postoperatively.

SUMMARY:
The sternotomy site is the most painful site after cardiac surgery. Local infiltration of ropivacaine through the multihole catheters in the bilaterosternal position (BLS) after sternotomy significantly reduces pain at rest and during mobilization, reduces opioids consumption, decreases postoperative complications, improves patient comfort and satisfaction and reduced hospital costs. In this study our hypothesis is to test the efficacity of local anesthetic administration via the catheters in the BLS position placed before the surgical incision.

DETAILED DESCRIPTION:
Goal of the study: Evaluation of the effectiveness of BLS technique on a composite endpoint (pain at rest, pain during patient mobilization and opioid consumption).

Open trial, therapeutic, prospective, monocentric. One group of patients who will benefits from the placement of two multihole catheters in BLS position:

* The ropivacaine group (40 patients): placement by the surgeon of two catheters in BLS position before the surgical incision. Administration of a bolus dose of 10 ml of ropivacaine 7, 5 mg/mL in each catheter followed by a continuous infusion of ropivacaine 2 mg/ml in a rate of 3 mL/h during the first 48 hours postoperatively.
* The control group (80 patients) from the two previous studies who underwent standard analgesia with PCA morphine.

ELIGIBILITY:
Inclusion Criteria:

* Patients who undergo scheduled cardiac surgery with sternotomy: aortic or mitral valve replacement, biological or mechanical, coronary bypass surgery
* Age under 85 years
* Patients who have given their consent according to the methods described in Title II of the book of the first Public Health Code
* Possession of Social Security insurance.

Exclusion Criteria:

* Emergency surgery
* Approach by thoracotomy
* Heart transplant
* Aortic dissection
* Redo surgery.
* Pregnant women
* Refusal of the protocol
* Protected minors or adults
* Pre-existing psychiatric pathology including known states of opioid addiction
* Long-term opioid medication
* Physical or intellectual inability to use a PCA
* Severe heart failure (ejection fraction less than 40% or PAH > 50 mmHg)
* Preoperative cardiogenic shock
* Severe preoperative chronic or acute renal failure with a creatinine clearance of less than 30 mL / min according to Cockroft's formula
* Known hypersensitivity to local anesthetics or to any component of the catheter
* Known allergy or hypersensitivity to any of the study drugs or analgesia protocol (ropivacaine, paracetamol, opiates).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2021-01-12 (Actual); Study Completion 2021-07-12 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | Day 2 postoperatively.
  The technique is considered as a fail if : pain rest > 3.5 /10 (0 = no pain; 10 maximum pain) or pain during mobilization > 3.5/10 (0 = no pain; 10 maximum pain)
Opioid consumption | Day 2 postoperatively.
  The technique is considered as a fail if morphine consumption > 35 mg

SECONDARY OUTCOMES:
ICU length of stay | Up to 6 months
  Days of ICU and hospital stay
Hospital length of stay | Up to 6 months
  Days of ICU and hospital stay
Patient satisfaction | Day 2 postoperatively.
  Patient satisfaction evaluation from the patient based on a simple Likert scale:
  0 = very bad; 1 = bad; 2 = medium; 3 = good; 4 = excellent.
Postoperative nausea and vomiting | Day 1 and 2 postoperatively.
  assessed by the Wengritzky intensity scale (if total score > 50, the nausea and vomiting are clincally significant)
Respiratory complications | Up to 6 months
  Occurrence of postoperative respiratory complications
Cardiac complications | Up to 6 months
  Occurrence of postoperative cardiac complications
Neurological complications | Up to 6 months
  Occurrence of postoperative neurological complications
Renal,complications | Up to 6 months
  Occurrence of postoperative renal complications
Infectious complications | Up to 6 months
  Occurrence of postoperative infectious complications
Chronic pain evaluation | Assessed at the 6th postoperative month
  Chronic pain assessed at the 6th postoperative month by DN4 (Neuropathic Pain Diagnostic 4) score

CONTACTS AND LOCATIONS:
Overall Officials: Vedat Eljezi, Dr, Principal Investigator — Pôle Anesthésie Réanimation / Service de Chirurgie Cardio-Vasculaire
Locations (1):
- CHU Clermont-Ferrand - Service de Chirurgie Cardio-Vasculaire, Clermont-Ferrand, Puy De Dôme, France